CLINICAL TRIAL: NCT02387281
Title: Freezing of Gait: Clinical, Cognitive, and Imaging Features
Acronym: FOG
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Stewart Factor, Professor, Emory University
Other Study IDs: IRB00073518
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- PD with FOG "on": Subjects diagnosed with Parkinson disease (PD) and sub-categorized as "on" freezing of gait (FOG) based on evaluation using motion capture
- PD with FOG "off": Subjects diagnosed with Parkinson disease (PD) and sub-categorized as "off" freezing of gait (FOG) based on evaluation using motion capture
- PD without FOG: Subjects with Parkinson disease (PD) and an absence of freezing of gait (FOG)
- Non-PD with FOG: Subjects with freezing of gait (FOG) and an absence of Parkinson disease (PD) (exception granted for those with FOG and atypical parkinsonism: PSP or MSA)

SUMMARY:
Freezing of gait (FOG) is among the most disabling motor features of Parkinson disease (PD) and is present in other forms of parkinsonism as well. FOG is a brief (usually lasting <30 seconds) episode of absence or a greatly reduced forward movement of the feet despite intention to walk. It typically occurs when patients initiate gait (so-called "start hesitation") and when attempting to turn. It is a leading cause of falls and often results in a wheelchair-dependent state. FOG greatly interferes with activities of daily living, causes social isolation and poor quality of life.

FOG is one of the least understood features of PD. It possibly may develop independent of the other motor features of the disease, and be caused by specific pathological changes in the brain. Previous studies on FOG have shown conflicting information and have not lead to clear understanding of the pathophysiology. One key reason for this is that there appears to be multiple subtypes which have rarely been taken into account.

The purpose of this study is to show that different types of FOG exist and to see if there is a connection to cognitive differences or gait patterns.

DETAILED DESCRIPTION:
This study is an observational study to assess FOG via using multiple methods such as: clinical features, imaging, cognition and dopamine blood levels. The study consists of four parts (plus an optional fifth part) that will be completed over two-three separate days within a 30 day span. The four parts will not necessarily be performed in this order. Part one will be clinical and written questionnaire assessments of PD and FOG followed by 3D motion capture evaluations. Part two are cognitive or neuropsychiatric assessments. Part three is a magnetic resonance image (MRI) to examine the brain structure. Part four is Positron Emission Tomography (PET) imaging scan that measures norepinephrine transporter levels. The optional part 5 is a lumbar puncture that will measure cerebrospinal fluid catecholamines and proteomics.

ELIGIBILITY:
Inclusion Criteria for Parkinson disease (PD) subjects with freezing of gait (FOG):

* Diagnosis of PD by United Kingdom Brain bank criteria
* Hoehn & Yahr stage I-IV
* Levodopa treated and responsive
* Able to manage 12 hours off dopaminergic medication
* Age 18-85 years
* Presence of FOG by history and seen by examiner at their clinical office visit or in a video taken at home
* Able sign a consent document and willing to participate in all aspects of the study
* Able to have an MRI scan (no pacemakers or history of claustrophobia)

Exclusion Criteria for Parkinson disease (PD) subjects with freezing of gait (FOG):

* Dementia that precludes completing study protocol
* Stage V PD - unable to walk independently when "off"
* History of FOG without ever being seen to have it
* Atypical parkinsonism: Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD), Vascular Parkinsonism
* Treatment with medications that cause parkinsonism: drug-induced parkinsonism
* Any neurological or orthopedic disorders that interfere with gait
* Treatment with medications that will interfere with NET-PET (norepinephrine transporter-positron emission tomography) ligand binding

  a. Noradrenergic drugs: methylphenidate, atomoxetine, serotonin-norepinephrine reuptake inhibitors (e.g., venlafaxine)
* Absence or loss of levodopa response
* Any contraindications for MRI scan including pacemaker, deep brain stimulator, bladder stimulator, etc.

Inclusion Criteria for Parkinson disease (PD) subjects but no freezing of gait (FOG):

* Diagnosis of PD by United Kingdom Brain bank criteria
* Hoehn & Yahr stage I-IV
* Levodopa treated and responsive
* Able to manage 12 hours off dopaminergic medication
* Age 18-85 years, age, gender and duration matched to the PD with FOG recruits
* Absence of FOG by history and by exam, confirmed by caregiver and FOG-Q item 3 score of 0.
* Able sign a consent document and willing to participate in all aspects of the study
* Able to have an MRI scan (no pacemakers or history of claustrophobia)

Exclusion Criteria for Parkinson disease (PD) subjects but no freezing of gait (FOG):

* Dementia that precludes completing study protocol
* Stage V PD - unable to walk independently when off.
* History of FOG at any time
* Atypical parkinsonism: Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD), Vascular Parkinsonism
* Treatment with medications that cause parkinsonism: drug-induced parkinsonism
* Any neurological or orthopedic disorders that interfere with gait
* Treatment with medications that will interfere with NET-PET ligand binding
* Absence or loss of levodopa response
* Any contraindications for MRI scan including pacemaker, deep brain stimulator, bladder stimulator, etc.

Inclusion Criteria for subjects with freezing of gait (FOG) but not Parkinson disease (PD):

* Diagnosis of Primary Progressive Freezing gait by accepted Criteria 71
* Diagnosis of atypical parkinsonism; Progressive Supranuclear Palsy (PSP) or Multiple System Atrophy (MSA) with predominant and early onset FOG.
* Hoehn & Yahr Stage I-IV parkinsonism
* Limited response to Levodopa but FOG unresponsive, but may be on levodopa or other dopaminergic medications
* Age 18-85 years
* Presence of FOG by history and seen by examiner at their clinical office visit or in a video taken at home
* MRI scan demonstrating no structural lesions: stroke, tumor or hydrocephalous
* Able sign a consent document and willing to participate in all aspects of the study
* Able to have an MRI scan (no pacemakers or history of claustrophobia).

Exclusion Criteria for subjects with freezing of gait (FOG) but not Parkinson disease (PD):

* Dementia that precludes completing study protocol
* Stage V Parkinsonism - unable to walk independently.
* Treatment with medications that cause parkinsonism: drug-induced parkinsonism
* MRI scan demonstrating structural lesions or hydrocephalous
* Notable levodopa response suggesting a diagnosis of PD including motor fluctuations or dyskinesia.
* Any neurological or orthopedic disorders that interfere with gait.
* Treatment with medications that will interfere with NET-PET ligand binding.
* Any contraindications for MRI scan including pacemaker, deep brain stimulator, bladder stimulator, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Freezing of gait (FOG) patients with Parkinson disease (PD) will be selected from the Emory Movement Disorders Center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | Baseline
  MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The Part III motor examination has 18 items, which are rated from 0-4, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
Response to levodopa | Baseline
  Subjects will be assessed in the "on" and "off" states to classify them properly according to pharmacological response to levodopa
Classification of FOG using motion capture | Baseline
  Classifying of FOG ("on" and "off") will be done measuring gait physiology though 3-dimensional motion capture between and during FOG episodes.
Plasma concentrations of levodopa | Baseline
  Levodopa plasma concentrations measured by modified high-performance liquid chromatography with electrochemical detection method during "on" and "off" episodes.

SECONDARY OUTCOMES:
Dot Counting task score | Baseline
  Dot counting is a verbal working memory task where the examinee looks at a computer screen with a mixed array of green circles, blue circles and blue squares, and instructed to count all of the blue circles on the screen one at a time and remember the final total. Once the examinee finishes counting the blue circles on one screen, the examiner switches the display to a different mixed array of green circles, blue circles and blue squares. The examinee is instructed to count the blue circles in the new display. The number of different displays presented to the examinee in each trial increases from two to seven over six trials. After counting the blue circles on all of the displays presented within a trial, the examinee recalls the total number of blue circles in each of the different displays in the order in which they were presented. The task includes six trials with possible scores ranging from 0 to 27.
N-back task score | Baseline
  The n-back paradigm is a widely used measure to assess spatial working memory. The 1-back requires maintaining and updating 1 location at a time. The examinee is shown a series of 2.4 cm white squares that appear in 15 different locations on a black computer screen. Each square is presented for 1000 ms. All of the locations are equidistant from the center of the screen. The 1-back consists of one block of 30 trials, ten of which match the location of the previous square, and 20 that are in a different location. Scoring is based on the number of accurate responses out of 30 trials.
Flanker task score | Baseline
  The Flanker task assesses an individual's ability to inhibit a prepotent response. A row of five arrows is presented in the center of the screen. The examinee is required to indicate whether the centrally presented arrow is pointing either to the left or right by pressing the left or right arrow key. The examinee is presented with two different conditions during the task, incongruent and congruent. In the congruent trials, the non-target arrows point in the same direction as the target arrow and in the incongruent trials they point in the opposite direction.The stimuli are presented in a random order with each condition being presented 24 times resulting in 48 total trials. Scoring is based on the number of accurate responses out of 48 trials.
Dimensional Set Shifting task score | Baseline
  The Dimensional Set Shifting task requires the individual to alternate between responding to shape vs. color of stimuli. Examinees are required to match a stimulus on the top of the screen to one of two stimuli in the lower corners of the screen. In task-homogeneous blocks, participants perform either Task A (e.g., classifying shapes) or Task B (e.g., classifying colors). In task-heterogeneous blocks, participants alternate between the two tasks pseudo-randomly. The combination of task-homogeneous and task-heterogeneous blocks allows measurement of general switch costs (latency differences between heterogeneous and homogeneous blocks) and specific switch costs (differences between switch and non-switch trials within the heterogeneous block). Scoring is based on the number of accurate responses out of 104 trials.
Digit Span Test score | Baseline
  The digit span test forward assesses attention and short-term memory. The digit span test backward assesses measures working memory. For the forward test, the examinee is told to listen carefully because the examiner will say a series of numbers and ask him/her to repeat them back to in the same order. For the backward test, the examiner will ask the examinee to repeat the numbers backwards, that is, by starting with the last number said and going backwards to the first number said. This process continues until the examinee can no longer remember either the full sequence of numbers or the correct order. Both forward and reverse trials are given twice. The Digit Span test is scored by the amount of numbers the examinee was able to remember in each test. The examiner must add the total number of correct sequences, backwards and forwards.
Number of seconds required to complete Trail Making Test (TMT): Trails A and Trails B | Baseline
  Trail A assesses scanning ability and psychomotor speed. Trail B assesses executive function. In Part A, the circles are numbered 1 - 25, and the participant should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the participant draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The participant should be instructed to connect the circles as quickly as possible. The participant is timed as he or she connects the "trail." If the participant makes an error, point it out and allow the participant to correct it. Errors affect the participant's score only in that the correction of errors is included in the completion time for the task. Participants are scored by the number of seconds taken to complete the task, with high scores revealing greater impairment.
Wisconsin Card Sorting Test (WCST) score | Baseline
  The WCST measures cognitive flexibility and problem solving skills. The WCST consists of a pack of 4 stimulus cards and 48 response cards which are devised so that each card contains from 1 to 4 identical figures of a single color. Individually administered, it requires the participant to sort the cards according to different principles (ie, by color, form, or number). As the test progresses, there are unannounced shifts in the sorting principle which require the participant to alter his or her approach.The 'number of categories' measures the number of correct responses. The percentage of perseverative errors provides the concentration of perseverative errors in relation to the overall test performance.
Brief Visuospatial Memory Test score | Baseline
  Brief Visuospatial Memory Test (BVMT) is a measure of visuospatial memory. This task includes three trials of six geometric figures printed on separate pages. The participant views the stimulus page for 10 seconds and is asked to draw as many of the figures as possible in their correct location on a paget. A Delayed Recall Trial is administered after a 30-minute delay. Scoring is based on accuracy of the figure as well as its location on the page. A range of 0-12 per trial is possible (0-36 total). Higher scores are better.
Hopkins Verbal Memory Test Total Recall score | Baseline
  Hopkins Verbal Learning Test (HVLT) provides a brief assessment of immediate recall. It is administered by reading the words aloud, then asking the participant to verbally repeat the list of words (immediately), and identify the words from a word list that is presented verbally. The participant is read a list of 12 words and is then asked to recall as many of the words as possible. Tasks include three learning trials, which, when combined produce a total recall score.The HVLT total recall score ranges from 0 to 36 with 36 being the highest and best possible score.
Hopkins Verbal Memory Test Delayed Recall score | Baseline
  Hopkins Verbal Learning Test (HVLT) provides a brief assessment of delay recall. It is administered by reading the words aloud, then asking the participant to verbally repeat the list of words (after a 20-25 minute delay), and identify the words from a word list that is presented verbally. The participant is read a list of 12 words and is then asked to recall as many of the words as possible. The HVLT delayed recall score ranges from 0 to 12 with 12 being the highest and best possible score.
Number of correct trials in Morris Water Maze Paradigm | Baseline
  Morris Water Maze (MWM) Paradigm is used to study spatial memory and learning. The MWM is a virtual water maze paradigm in which the hidden platform is continually re-located. The participant has to locate a hidden platform to escape the water. The number of correct trials will be the score.
Number of correct trials in Recognition of Scenes | Baseline
  Recognition of Scenes is used to assess emotional memory. The Recognition of Scenes task requires the participant to recall various scenes that have different emotional valences. The number of correct trials will be the score.
Number of correct responses for Confrontation Naming task | Baseline
  Confrontation naming tasks are used to assess impairments of word-finding abilities in individuals with various types of neurologic impairments. Confrontation naming involves the selection of a specific label corresponding to a viewed stimulus, usually a picture, of a viewed object or action. The number of correct responses will be the score.
Verbal Fluency in Naming Categories | Baseline
  Fluency is measured by timed word retrieval. Participants are given 60 seconds to name as many words as possible within a given category. The more words named, the better cognition
Benton Judgment of Line Orientation Test | Baseline
  Line orientation assesses spatial perception and orientation without requiring a motor output. The Benton Judgment of Line Orientation Test measures a person's ability to match the angle and orientation of lines in space. Participants are asked to match two angled lines to a set of 11 lines that are arranged in a semicircle and separated 18 degrees from each other.The test is a standardized test with 30 items with the minimum score being 0, indicating low visual spatial cognition and the maximum score being 30, indicating high visual spatial cognition.
Number of correct responses for Mental Rotation Task | Baseline
  Mental rotation is the ability to rotate mental representations of two-dimensional and three-dimensional objects as it is related to the visual representation of such rotation within the human mind.In a mental rotation test, the participant is asked to compare two 3D objects (or letters), often rotated in some axis, and state if they are the same image or if they are mirror images (enantiomorphs). Commonly, the test will have pairs of images each rotated a specific amount of degrees (e.g. 0°, 60°, 120° or 180°). Some pairs will be the same image rotated, and others will be mirrored. The participant will be shown a set number of the pairs. The participant will be scored on how accurately they can distinguish between the mirrored and non-mirrored pairs. The number of correct responses will be the score.
Scale for the Assessment of Positive Symptoms (SAPS) score | Baseline
  Scale for the Assessment of Positive Symptoms (SAPS) assesses the presence of psychotic symptoms. There are 34 items rated on a scale of 0-5 with 0=none and 5=severe for a minimum score of 0 and a maximum score of 170. There are 4 subscales: Hallucinations (minimum score 0; maximum score 35); Delusions (minimum score 0; maximum score 65); Bizarre Behavior (minimum score 0; maximum score 25); Positive Formal Thought Disorder (minimum score 0; maximum score 45). Each subscale contains one additional question as a Global Rating - or overall measure for that particular subscale. The sum of these questions constitutes the Total Global Score (minimum 0, maximum 20). The values for the Global items are included in the Total Composite score. In each case, the higher the score, the greater the severity of symptoms.
Beck Depression Inventory (BDI) score | Baseline
  Beck Depression Inventory (BDI) is a self-report rating inventory measuring characteristic attitudes and symptoms of depression consisting of 21 items with each item rated on a four point scale (0=not present to 3=severe). The accepted ranges are as follows: 0 to 9 indicates no depression, 10 to 18 indicates mild to moderate depression, 19 to 29 indicates moderate to severe depression and 30 to 63 indicates severe depression.
Beck Anxiety Inventory (BAI) score | Baseline
  Beck Anxiety Inventory (BAI) is a self-report rating inventory measuring general anxiety consisting of 21 items with each item rated on a four point scale (0=not present to 3=severe). Scores range from 0-63, with higher scores indicating greater anxiety.
Questionnaire for Impulsive-Compulsive disorders in Parkinson's disease (QUIP) | Baseline
  Questionnaire for Impulsive-Compulsive disorders in Parkinson's disease (QUIP) is a rating scale designed to measure severity of symptoms and support a diagnosis of impulse control disorders and related disorders in Parkinson's disease. QUIP has four primary questions (pertaining to commonly reported thoughts, urges/desires, and behaviors associated with Impulse control disorders (ICDs)), each applied to the 4 ICDs (compulsive gambling, buying, eating, and sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). It uses a 5-point Likert scale (score 0-4 for each question) to gauge the frequency of behaviors. Scores for each ICD and related disorder range from 0 to 16, with a higher score indicating greater severity (ie, frequency) of symptoms. The total QUIP score for all ICDs and related disorders combined ranges from 0 to 112.
New Freezing of Gait Questionnaire (NFOG-Q) score | Baseline
  The NFOG-Q is used to quantify FOG severity and frequency in the daily living. It is a self-report measure that begins with the presentation of a short video to illustrate FOG during walking, turning and starting gait and then follows with questions related to frequency and duration of each type of FOG episode. Part I detects the presence of FOG using a dichotomous item in which individuals are classified as a freezer (FR) or a non-freezer (NFR). Parts II and III are designed for FRs only, providing a total summed score between 0 and 28. Part II (items 2-6, scoring range 0-19) rated the severity of FOG based on its duration and frequency. Part III rates the impact of FOG on daily life (items 7-9, scoring range 0-9).
Measurement of neuromelanin-containing neurons in the locus ceruleus and substantia nigra | Baseline
  The high-resolution neuromelanin images using a magnetic resonance imaging (MRI) technique will examine noradrenergic neurons in the brain.
Measurement of norepinephrine transporter levels | Baseline
  Positron emission tomography (PET) is a technique for measuring the 3-dimensional distribution of radioactive tracers in the living human. The norepinephrine transporter (NET) ligand, [11C]MeNER, with PET imaging will measure changes in norepinephrine terminals in key brain regions and compare FOG subtypes and non-FOG PD.
Cerebrospinal fluid (CSF) biomarkers | Baseline
  Cerebrospinal fluid (CSF) collected via lumbar puncture to measure catecholamines and proteomics.
Montreal Cognitive Assessment (MoCA) score | Baseline
  The Montreal Cognitive Assessment (MoCA) is a brief 30-point screening instrument that identifies subjects with mild cognitive impairment. Total MoCA score represents the sum of these 30-points, with a lower score indicating greater cognitive impairment. 30 is the maximum score, with a score of 26 or higher considered normal and below 26 indicative of Mild Cognitive Impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Factor, DO, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Movement Disorders Center, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia